CLINICAL TRIAL: NCT04830813
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter Phase 3 Clinical Study of Chiauranib Capsule in Patients With Progressed or Relapsed Small-cell Lung Cancer After 2 Lines Chemotherapy (CHIS)
Brief Title: Phase 3 Clinical Study of Chiauranib Capsule in Patients With Small-cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chipscreen Biosciences, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAR302
Record Dates: First submitted 2021-03-29; First posted 2021-04-05 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-11

CONDITIONS: Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — chiauranib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chiauranib (Experimental): Patients take Chiauranib capsules 50mg, orally once daily, 21 days as a cycle until objective disease progression.
  Interventions: Drug: Chiauranib
- Placebo (Placebo Comparator): Participants received Chiauranib placebo capsule matching Chiauranib orally once daily until objective disease progression.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Chiauranib — Patients take Chiauranib capsules 50mg, orally once daily, 21 days as a cycle until objective disease progression.
  Other Names: CS2164
  Arms: Chiauranib
Drug: Placebo — Participants received Chiauranib placebo capsule matching Chiauranib orally once daily until objective disease progression.
  Other Names: Simulation tablet of Chiauranib
  Arms: Placebo

SUMMARY:
Chiauranib , which simultaneously targets against VEGFR/Aurora B/CSF-1R, several key kinases involved in tumor angiogenesis, tumor cell mitosis, and chronic inflammatory microenvironment.

DETAILED DESCRIPTION:
Chiauranib is a novel orally active multi-target inhibitor that simultaneously inhibits the angiogenesis-related kinases (VEGFR2, VEGFR1, VEGFR3, PDGFRa and c-Kit), mitosis-related kinase Aurora B and chronic inflammationrelated kinase CSF-1R in a high potency manner with the IC50 at a single-digit nanomolar range. In particular, Chiauranib showed very high selectivity in the kinase inhibition profile with little activity on off-target non-receptor kinases, proteins, GPCR and ion channels, indicative of a better drug safety profile in terms of clinical relevance.

In July 2017, the sponsor initiated a phase Ib/II trial (CAR105). As of October 9, 2020, a total of 42 subjects entered the safety analysis and 41 subjects entered the efficacy analysis. The results of the phased trial analysis show the preliminary efficacy of this product in the treatment of SCLC at ≥3 lines.

This clinical trial is studying the efficacy and safety of chiauranib works in treating patients with relapsed or refractory small cell lung cancer, in the meantime, exploreing the latent biomarkers accompany with chiauranib, as well as the relevancy of which and clinical benefit.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age ≥ 18 years and ≤75 years;
* Cytologically or histologically confirmed small cell lung cancer;
* Patients have received at least 2 different systemic chemotherapy regimens (contained platinum based regimen) , and progressed or relapsed
* At least one measurable lesion that can be accurately assessed ( RECIST1.1 criteria). If the only site of measurable disease is in a previously irradiated area, the patient must have documented progression of disease in this area.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
* Laboratory criteria are as follows:

  * Complete blood count: absolute neutrophil count (ANC) ≥1.5×10^9/L ; platelets ≥75×10^9/L; hemoglobin (Hb) ≥80g/L ;
  * Biochemistry test: total bilirubin≤1.5×ULN; alanine aminotransferase (ALT) , aspartate aminotransferase(AST)≤2.5×ULN(ALT,AST≦5×ULN if liver involved); serum creatinine(cr)≤1.5×ULN;
  * Coagulation test: International Normalized Ratio (INR) < 1.5.
* Life expectancy of at least 3 months.
* All patients must have given signed, informed consent prior to registration on study.

Exclusion Criteria:

* Patients who known to brain metastases with neurological symptoms;
* Screening period imaging shows that the tumor has invaded the periphery of important blood vessels or the investigator judges that the tumor is likely to invade important blood vessels and cause hemorrhage during the trial
* Pleural fluid, ascites, pericardial effusion with clinical symptoms or need to be drained during the screening period
* Patients with second primary cancer, except: adequately treated basal cell or squamous cell skin cancer, curatively treated in-situ cancer of the cervix, unless received curative treatment and with documented evidence of no recurrence during the past five years
* Patients who have been used aurora kinase inhibitors, or VEGF/VEGFR inhibitors
* Patients have used any anti-cancer therapy, including adiotherapy, chemotherapy, immunotherapy, target therapy, and other anti-tumor treatments within 28 days before the first dose
* Patients have used experimental drugs or devices within 28 days before the first dose
* Patients received major surgical operations within 28 days before the first dose, or patients with serious non-healing wounds, ulcer or fracture at the time of screening
* With the exception of alopecia, any ongoing toxicities (>CTCAE grade 1) caused by previous cancer therapy
* Patients with uncontrolled or significant cardiovascular disease, including:

  * Grade II or higher Congestive heart failure, unstable angina pectoris, myocardial infarction (NYHA Classification) within 6 months prior to study entry; or arrhythmia requiring treatment, or Left Ventricular Ejection Fraction (LVEF) < 50% during screening stage.
  * Primary cardiomyopathy (dilated cardiomyopathy, hypertrophic cardiomyocyte, arrhythmogenic right ventricular cardiomyopathy, restrictive cardiomyopathy, et,al).
  * History of significant QT interval prolongation, or Corrected QT Interval QTc≥450ms(male),QTc≥470ms（female）at screening.
  * patient's treatment record of using at least 2 antihypertensive drugs at the same Within 14 days before the first dose, or uncontrolled hypertension (> 140/90 mmHg) during the screening period.
* Obstructive atelectasis that requires chest radiotherapy or surgery during the screening period or CT or MRI of the chest during the screening period shows interstitial lung disease or pulmonary fibrosis or lung inflammation that requires treatment, or within 6 months before the first dose history of pneumonia requiring oral or intravenous steroid treatment
* Patients with factors that could affect oral medication (such as dysphagia，chronic diarrhea, intestinal obstruction, After small bowel resection,etc), or undergone gastrectomy, or history of gastrointestinal perforation
* Proteinuria positive(≥1g/24h)
* Active bleeding within 2 months before the first dose, or anticoagulant drugs are being taken during the screening period, or the investigator judges that there is a high risk of bleeding during the screening period
* History of deep vein thrombosis or pulmonary embolism within 6 months before the first dose
* Active infections that require systemic treatment (oral, intravenous infusion) during the screening period
* Screening for HIV antibody positive
* Screening test for hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) positive with virus replication, hepatitis C antibody (HCV-Ab) positive with virus replication
* Any mental or cognitive disorder, that would impair the ability to understand the informed consent document, or the compliance of study
* Candidates with drug and alcohol abuse
* Women of childbearing potential not willing to use and utilize an adequate method of contraception (such as intrauterine device, contraceptive and condom) throughout treatment and for at least 12 weeks after the last dose; pregnant or breastfeeding women; the result of urine pregnancy test was positive at screening; Man participants not willing to use and utilize an adequate method of contraception throughout treatment.
* Any other condition which is inappropriate for the study according to investigators' judgment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2021-03-05 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
PFS | From date of the first dose of study drug until the date of first documented progression or relapse or date of death from any cause, whichever came first, assessed up to 24 months
  Progression-free survival
OS | From date of the first dose of study drug until the date of death from any cause, assessed up to 24 months
  Overall survival

SECONDARY OUTCOMES:
ORR | Up to a minimum 24 weeks after the last participant's first dose, or progression, or 75% subjects died
  Objective reponse rate
DOR | from the date of first documented objective response until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  Duration of response
DCR | Up to a minimum 24 weeks after the last participant's first dose, or progression, or 75% subjects died
  Disease-control rate
percentage of AEs | 28 days after the last participant 's last medication or new anti-tumor therapy
  Safety

CONTACTS AND LOCATIONS:
Overall Officials: Yuankai Shi, Principal Investigator — Cancer Hospital,Chinese Academy of Medical Sciences and Peking Union Medical College
Locations (1):
- Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No